CLINICAL TRIAL: NCT06455527
Title: HRV-Guided tDCS: Integrating A Biomarker For Clinical Utility
Brief Title: Heart Rate Variability (HRV)-Guided Transcranial Direct Current Stimulation (tDCS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 24-00536
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Depression
Keywords: Depression; Heart Rate; tDCS; Brain stimulation; telehealth
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): Participants randomized to the Active tDCS arm will complete 10 sessions of 30-minute active remotely supervised (RS)-tDCS with chest strap and impedance-based HRV data collection over the course of approximately 2-4 weeks.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Participants randomized to the Active tDCS arm will complete 10 sessions of 30-minute sham RS-tDCS with chest strap and impedance-based HRV data collection over the course of approximately 2-4 weeks.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — tDCS will be delivered using the 1x1 Mini CT tDCS device. For active tDCS, the device is programmed to ramp up to 2.0 mA (for 30 seconds), provide constant current throughout the session (29 minutes), and then ramp down (for 30 seconds) at the end. Participants will receive 10 sessions of tDCS over the course of this study on weekdays (M-F).
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Sham tDCS will be delivered using the 1x1 Mini CT tDCS device. For sham tDCS, the device is programmed to ramp up to 2.0 mA (for 30 seconds) followed by a ramp down (30 seconds), with no current delivery for 28 minutes, and then ramp up (for 30 seconds) and down (for 30 seconds) at the end. Participants will receive 10 sessions of sham tDCS over the course of this study on weekdays (M-F).
  Arms: Sham tDCS

SUMMARY:
This technology development project will be informed and guided by initial data collection of human subject data. For this purpose, the investigators will recruit n=100 people with mild to moderate depression in a double-blinded, parallel-arm, sham-controlled data collection period administered at home and using the investigator's remotely supervised (RS) tDCS protocol. Enrolled participants will complete 10 days of 30-minute tDCS (2.0, DLPFC left anodal) using the RS-tDCS protocol. During each daily session, standard HR and impedance-based HR (i-HR), obtained from the tDCS headset, will be collected to identify a possible marker of response to tDCS in depression. Participants will be randomized 2:1 to active vs. sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate depression (Beck Depression Inventory(BDI)-II 14-28)
* Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-V-TR) Depressive episode
* Wide Range Achievement Test (WRAT)-4th Reading Recognition subtest standard score >85

Exclusion Criteria:

* Primary neurologic, psychiatric (e.g., multiple sclerosis, stroke, Parkinson's disease, spinal cord injury, intracranial mass, traumatic brain injury (TBI), epilepsy, mild cognitive impairment (MCI), or dementia), or major medical disorder (e.g., history of myocardial infarction, diabetes, thyroid disease, arrhythmia, atrial fibrillation) (medical history review)
* DSM-V-TR bipolar depression, psychotic disorder, or alcohol or substance use disorder (M.I.N.I.)
* Active or high suicidality risk (Columbia-Suicide Severity Rating Scale, C-SSRS), or otherwise judged as inappropriate by the study clinicians
* History of a heart transplant, presence of permanent pacemaker implant or Left Ventricular Assist Device
* Use of certain medications that can affect heart rate variability, such as beta-blockers, calcium channel blockers, or cardiac glycosides
* Use of antidepressant, antipsychotic, anxiolytic, or stimulant medications
* Pregnant or planning pregnancy during the study period
* Seizure disorder or recent (<5 years) seizure history
* Presence of metal objects in the head/neck
* Any skin disorder or skin sensitive area near stimulation locations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Average Heart Rate (HR) Measured Using Polar H10 Chest Monitor | Up to Week 4
  HR will be measured using Polar H10 Chest Monitor at each daily tDCS session.
Average HR Measured Using i-HR Data Logger | Up to Week 4
  HR will be measured using an impedance-based HR (i-HR) data logger attached to the Mini-CT tDCS device at each daily tDCS session.

SECONDARY OUTCOMES:
Change in Montgomery Ӓsberg Depression Rating Scale (MADRS) Score | Baseline, End of Intervention (Up to Week 4)
  MADRS is a 10-item assessment of severity of depressive episodes in patients with mood disorders. Each item is rated on a scale from 0-6. The total score is the sum of responses and ranges from 0-60; higher scores indicate greater severity of depressive episodes.
Change in State-Trait Anxiety Inventory for Adults (STAI): State Score | Baseline, End of Intervention (Up to Week 4)
  STAI is a 40-item questionnaire measuring state and trait anxiety. Each item is rated on a 4-point Likert scale. The range of possible scores for state anxiety ranges from a minimum score of 20 to a maximum score of 80; higher scores indicate greater state anxiety.
Change in State-Trait Anxiety Inventory for Adults (STAI): Trait Score | Baseline, End of Intervention (Up to Week 4)
  STAI is a 40-item questionnaire measuring state and trait anxiety. Each item is rated on a 4-point Likert scale. The range of possible scores for trait anxiety ranges from a minimum score of 20 to a maximum score of 80; higher scores indicate greater trait anxiety.
Change in Positive and Negative Affect Schedule (PANAS-SF): Positive Affect Score | Baseline, End of Intervention (Up to Week 4)
  PANAS-SF is a self-report questionnaire that consists of two 10-item scales (20 items total) to measure both positive and negative affect. Each item is rated on a scale from 1 (very slightly or not at all) to 5 (extremely). The total positive affect score is the sum of affect item responses and ranges from 10 - 50; higher scores represent higher levels of positive affect.
Change in Positive and Negative Affect Schedule (PANAS-SF): Negative Affect Score | Baseline, End of Intervention (Up to Week 4)
  PANAS-SF is a self-report questionnaire that consists of two 10-item scales (20 items total) to measure both positive and negative affect. Each item is rated on a scale from 1 (very slightly or not at all) to 5 (extremely). The total negative affect score is the sum of negative item responses and ranges from 10 - 50; lower scores represent lower levels of negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Pilloni, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Giuseppina.Pilloni@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposes to use the data will be granted access upon reasonable request. Requests should be directed to Giuseppina.Pilloni@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.